CLINICAL TRIAL: NCT00728403
Title: Long Term Metabolic and Therapeutic Effects of Combined Treatment of American Ginseng (Panax Quinquefolius L.) Extract and Korean Red Ginseng (Steamed Panax C.A. Meyer) Extract in the Treatment of Type 2 Diabetes
Brief Title: Metabolic and Therapeutic Effects of American and Korean Red Ginseng in the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122380
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Asian ginseng; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): American Ginseng and American Red Ginseng Capsules
  Interventions: Dietary Supplement: American Ginseng (Panax quinquefolius L.) and Korean Red Ginseng (steamed Panax C.A. Meyer)
- 2 (Experimental): American Ginseng Capsules
  Interventions: Dietary Supplement: American Ginseng (Panax quinquefolius L.)
- 3 (Placebo Comparator): Placebo Capsules
  Interventions: Dietary Supplement: Wheat Bran

INTERVENTIONS:
Dietary Supplement: American Ginseng (Panax quinquefolius L.) and Korean Red Ginseng (steamed Panax C.A. Meyer) — 1.5 grams American Ginseng and 1.5 grams Korean Red Ginseng are to be taken in capsulated form. Two capsules are taken with every meal, for a total of 6 capsules per day for 12 weeks
  Arms: 1
Dietary Supplement: American Ginseng (Panax quinquefolius L.) — 3 grams of American Ginseng is to be taken in capsulated form. Two capsules are taken with every meal, for a total of 6 capsules per day for 12 weeks
  Arms: 2
Dietary Supplement: Wheat Bran — 3 grams of Wheat Bran is to be taken in capsulated form. Two capsules are taken with every meal, for a total of 6 capsules per day for 12 weeks
  Arms: 3

SUMMARY:
The study is a 2 phase double blind randomized placebo control trial. The objective is to asses the metabolic and therapeutic effects of American Ginseng (Panax quinquefolius L.) extract and Korean Red Ginseng (steamed Panax C.A. Meyer) extract in the management of type 2 diabetes in a 12 week period. One Hundred and twenty subjects with type 2 diabetes (hyperglycemia key inclusion criteria: HbAlc≥6.5% - ≤ 8.1% ) will participate in the study (36 men and 36 post-menopausal women).

ELIGIBILITY:
Inclusion Criteria:

* presence of type 2 diabetes (at least 1 year) as defined by A1c between ≥6.5% and ≤8.1%, at recruitment,
* treatment with diet or oral hypoglycemic medication be unchanged starting at least 2 months prior to the beginning of the study (at recruitment, week -8)
* between the age of 40 and 75 years
* systolic blood pressure <140 and diastolic blood pressure <90
* clinically euthyroid (measuring T3 and T4)
* normal renal and liver functions
* post-menopausal or non-pregnant women (Post-menopausal includes: those females with more than a year of cessation of menstruation)
* a negative result on a pregnancy test administered at screening
* subjects taking an effective form of birth control (example: condom, abstinence, etc.)
* willing to comply with the study protocol and sign a consent form

Exclusion Criteria:

* individuals with bleeding disorders
* individuals with allergies to nitroglycerin
* planned surgery, pregnancy or breastfeeding
* taking insulin; clinically significant diabetes complications (retinopathy, nephropathy, or neuropathy); serum triglycerides ≥ 4.5 mmol/L
* increased A1c level of more than 2% from baseline during the study
* history of angina or heart attack
* use of ginseng or any natural health products with glucose modulating and/or anti-platelet activity within 2 months
* BMI > 35 kg/m2 including a weight fluctuation of + 2kg during treatment periods
* smoke cigarettes; alcohol intake > 2 drinks/day
* the presence of any conditions which, in the opinion of the investigator, might jeopardize the health and safety of the subject or study personnel or adversely affect the study results, if the subject participated in the study
* Subjects taking Warfarin or Coumadin, prescription NSAIDs, chronic use of high-dose (>81mg) non-prescription NSAIDs, or selective serotonin reuptake inhibitors and monoamine oxidase inhibitors, or sympathomimetics or medications affecting nitric oxide levels, or any known or suspected sensitivity to any of the ingredients in the test product or placebo cannot participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
HbA1c levels and insulin sensitivity index using 3 different indices: ISI, HOMA, QUICKI | Weeks -4, 0, 6, 12

SECONDARY OUTCOMES:
Cholesterol, triglycerides, fasting & post-prandial blood glucose and insulin, C-reactive protein, lipid peroxidation, blood pressure, endothelial function, body fat composition | Weeks -4, 0, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Clinical Nutritian and Risk Factor Modification Centre; Alexandra Jenkins, PhD, Principal Investigator — Clinical Nutrition and Risk Factor Modificatrion Centre; Lawerence Leiter, MD, Principal Investigator — St. Michaels Hospital; Leanne De Souza, M.Sc., Principal Investigator — Clinical Nutrition and Risk Factor Modificatrion Centre
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada